CLINICAL TRIAL: NCT02258529
Title: A Phase 2, Single Arm Study Evaluating the Safety and Efficacy of Idelalisib in Combination With Rituximab for Previously Untreated Follicular Lymphoma and Small Lymphocytic Lymphoma
Brief Title: Idelalisib in Combination With Rituximab for Previously Untreated Follicular Lymphoma and Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-313-1414
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2017-04

CONDITIONS: Follicular Lymphoma; Small Lymphocytic Lymphoma
Keywords: Cancer; Indolent Non-Hodgkin Lymphoma; FL; SLL
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — idelalisib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idelalisib + rituximab (Experimental): Idelalisib + rituximab for up to 104 weeks
  Interventions: Drug: Idelalisib; Biological: Rituximab

INTERVENTIONS:
Drug: Idelalisib — 150 tablets administered orally twice daily
  Other Names: Zydelig®; GS-1101
Biological: Rituximab — 375 mg/m^2 administered intravenously (weekly for 4 weeks and then every 8 weeks from Week 12 up to Week 100)
  Other Names: Rituxan®; MabThera®

SUMMARY:
The primary objective of this study is to evaluate the overall response rate (ORR) and complete response (CR) rate to treatment with idelalisib in combination with rituximab in previously untreated adults with follicular lymphoma (FL) or small lymphocytic lymphoma (SLL).

An increased rate of deaths and serious adverse events (SAEs) among participants with front-line chronic lymphocytic leukemia (CLL) and early-line indolent non-Hodgkin lymphoma (iNHL) treated with idelalisib in combination with standard therapies was observed by the independent data monitoring committee (DMC) during regular review of 3 Gilead Phase 3 studies. Gilead reviewed the unblinded data and terminated those studies in agreement with the DMC recommendation and in consultation with the US Food and Drug Administration (FDA). All front-line studies of idelalisib, including this study, were also terminated.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of B-cell lymphoma
* No previous systemic treatment for lymphoma
* Subject demonstrates need for treatment for lymphoma
* Ann-Arbor Stage 2 (noncontiguous), 3, or 4 disease
* Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy
* Adequate performance status
* Required baseline laboratory data within protocol-specified parameters

Key Exclusion Criteria:

* Known history of transformed lymphoma or diffuse large cell lymphoid malignancy
* Known history of, or clinically apparent, central nervous system (CNS) lymphoma or leptomeningeal lymphoma
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of enrollment
* Known history of drug-induced liver injury, chronic active hepatitis B (HBV), chronic active hepatitis C (HCV), alcoholic liver disease, non-alcoholic steatohepatitis, cirrhosis of the liver, portal hypertension, primary biliary cirrhosis, or ongoing extrahepatic obstruction caused by cholelithiasis
* Ongoing inflammatory bowel disease
* Known human immunodeficiency virus (HIV) infection
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy, including systemic corticosteroids (> 10 mg prednisone or equivalent/day) with the exception of the use of topical, enteric, or inhaled corticosteroids as therapy for comorbid conditions and systemic steroids for autoimmune anemia and/or thrombocytopenia

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - Pacific Shores Medical Group, Long Beach, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - St. Agnes Hospital, Baltimore, Maryland
  - Prarie Lakes Health Care Systems, Inc., Watertown, South Dakota
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 14 September 2015. The last study visit occurred on 03 May 2016.
Pre-assignment Details: 20 participants were screened.
Groups:
- Idelalisib + Rituximab: Idelalisib (Zydelig®) 150 mg tablet twice daily for up to 104 weeks + rituximab 375 mg/m^2 intravenously (once weekly for 4 weeks and then every 8 weeks from Week 12 up to Week 100)
Period: Overall Study
Arm/Group | Idelalisib + Rituximab
Started | 10
Completed | 0
Not Completed | 10
Not completed — Study Terminated by Sponsor | 9
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set: all participants who received at least 1 dose of study drug.
Groups:
- Idelalisib + Rituximab: Idelalisib 150 mg tablet twice daily for up to 104 weeks + rituximab 375 mg/m^2 intravenously (once weekly for 4 weeks and then every 8 weeks from Week 12 up to Week 100)
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) was defined as the proportion of participants who achieve a confirmed complete or partial response during idelalisib treatment. ORR was to be assessed by an independent review committee (IRC).
Population: Due to the early termination of the study, efficacy data were not available for all participants, and therefore the prespecified analyses were not conducted.
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Safety Profile of Idelalisib as Measured by the Incidence of Adverse Events (AEs), Severe AEs (SAEs), AEs Leading to Idelalisib (IDL) Interruption, Idelalisib Dose Reduction, Premature Discontinuation of Idelalisib, or Death
Time Frame: Up to 24 weeks plus 30 days
Population: Intent-to-Treat (ITT) Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 10
percentage of participants
  Any AE | 90.0
  Any SAEs | 30.0
  Any AE Leading to Idelalisib Interruption | 60.0
  Any AE Leading to Idelalisib Dose Reduction | 30.0
  Any AE Leading to Premature Discontinuation of IDL | 10.0
  Any AE Leading to Death | 0

3. Secondary Outcome: Rate of Grade ≥ 3 Transaminase Elevations Based on Laboratory Findings
Description: The rate of Grade ≥ 3 transaminase elevations was defined as the number of participants with any Grade 3 or 4 alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevations.
Time Frame: Up to 24 weeks plus 30 days
Population: ITT Analysis Set: all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 10
percentage of participants
  Any Grade 3 or 4 ALT Elevation | 40.0
  Any Grade 3 or 4 AST Elevation | 10.0

4. Secondary Outcome: Idelalisib Trough and Peak Plasma Concentrations
Time Frame: Predose and 1.5 hour postdose at Weeks 2, 4, and 12
Population: Pharmacokinetic (PK) Analysis Set: all participants in the ITT Analysis Set who had the necessary baseline and on-study measurements to provide interpretable results for the specific parameters of interest.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 9
ng/mL
  Week 2 predose: number analyzed (Participants) | 8
  Week 2 predose | 216.2 (161.73)
  Week 2 1.5 hours postdose | 2240.0 (880.03)
  Week 4 predose: number analyzed (Participants) | 6
  Week 4 predose | 347.4 (365.57)
  Week 4 1.5 hours postdose: number analyzed (Participants) | 6
  Week 4 1.5 hours postdose | 2084.3 (1346.26)
  Week 12 predose: number analyzed (Participants) | 5
  Week 12 predose | 290.5 (373.08)
  Week 12 1.5 hours postdose: number analyzed (Participants) | 4
  Week 12 1.5 hours postdose | 1313.1 (1474.87)

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the the interval from the start of idelalisib treatment to the first documentation of complete or partial response.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the interval from the first documentation of complete response or partial response to the earlier of the first documentation of disease progression or death from any cause.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the interval from the start of idelalisib treatment to the earlier of the first documentation of disease progression or death from any cause.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval from enrollment to death from any cause.
Population: Due to the early termination of the study, efficacy data were not mature for all participants, and therefore the prespecified analyses were not conducted.
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

9. Secondary Outcome: Changes in Health-Related Quality of Life
Description: Changes in health-related quality of life was to be reported by participants using the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) questionnaire.
Population: Due to the early termination of the study, data were not available for all participants, and therefore this prespecified analysis was not conducted.
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (maximum: 24.1 weeks)
Description: ITT Analysis Set: all participants who received at least 1 dose of study drug.
Arm/Group | Idelalisib + Rituximab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=10)
Oedema peripheral (General disorders) | 1
Sepsis (Infections and infestations) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=10)
Neutropenia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ear pruritus (Ear and labyrinth disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 3
Mucosal inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 2
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatic steatosis (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Periportal oedema (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood cholesterol increased (Investigations) | 1
Liver function test increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, efficacy data were not available for all participants, and therefore the prespecified analyses were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years